CLINICAL TRIAL: NCT03511118
Title: Pharmacokinetics and Safety of Commonly Used Drugs in Lactating Women and Breastfed Infants
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: The Emmes Company, LLC (Industry); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Kanecia Obie Zimmerman, Associate Professor of Pediatrics, Duke University
Other Study IDs: Pro00088919; HHSN275201000003I/27500051 (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2018-04-23; First posted 2018-04-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lactating Women on Select DOI; Breastfed Infants of Mothers on Select DOI
MeSH Terms: interventions — Tranexamic Acid; Labetalol; Metformin; Nifedipine; Clindamycin; Oxycodone; Azithromycin; Escitalopram; Sertraline; Ondansetron; Ciprofloxacin; Doxycycline; Levofloxacin; Methylphenidate; Sumatriptan; Citalopram; cyclobenzaprine; Furosemide; Gabapentin; Hydrochlorothiazide; Hydroxyurea; Rosuvastatin Calcium; Topiramate; Trazodone; Valganciclovir; Venlafaxine Hydrochloride; Verapamil; remdesivir; Interleukin 1 Receptor Antagonist Protein; tocilizumab; Fluvoxamine; Amoxicillin; Bupropion; Duloxetine Hydrochloride; Hydrocodone; Levetiracetam; Paroxetine; Buprenorphine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leftover specimens will be sent to NICHD repository for unknown future use
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (38):
- Tranexamic acid (TXA): No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Tranexamic acid (TXA)
- labetalol: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: labetalol
- metformin: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: metformin
- nifedipine: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: nifedipine
- clindamycin: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: clindamycin
- oxycodone: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: oxycodone
- azithromycin: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: azithromycin
- escitalopram: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: escitalopram
- sertraline: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: sertraline
- ondansetron: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: ondansetron
- Ciprofloxacin: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Ciprofloxacin
- Doxycycline: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Doxycycline
- Levofloxacin: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Levofloxacin
- Methylphenidate: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Methylphenidate
- Sumatriptan: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Sumatriptan
- Citalopram: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Citalopram
- Cyclobenzaprine: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Cyclobenzaprine
- Furosemide: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Furosemide
- Gabapentin: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Gabapentin
- Hydrochlorothiazide: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Hydrochlorothiazide
- Hydroxyurea: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Hydroxyurea
- Rosuvastatin: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Rosuvastatin
- Topiramate: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Topiramate
- Trazodone: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Trazodone
- Valganciclovir: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Valganciclovir
- Venlafaxine: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Venlafaxine
- Verapamil: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Verapamil
- Remdesivir: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Remdesivir
- Anakinra: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Anakinra
- Tocilizumab: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Tocilizumab
- Fluvoxamine: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Fluvoxamine
- Amoxicillin: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Amoxicillin
- Bupropion: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Bupropion
- Buprenorphine: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Buprenorphine
- Hydrocodone: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Hydrocodone
- Levetiracetam: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Levetiracetam
- Paroxetine: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Paroxetine
- Duloxetine: No intervention, observational study and PK collections The study objectives are to characterize the PK and safety profile of DOIs that are commonly administered to lactating women.
  The primary focus of this analysis will be to determine drug concentrations in breastmilk and to estimate the relative infant dose.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Tranexamic acid (TXA) — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Tranexamic acid (TXA)
Drug: labetalol — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: labetalol
Drug: metformin — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: metformin
Drug: nifedipine — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: nifedipine
Drug: clindamycin — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: clindamycin
Drug: oxycodone — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: oxycodone
Drug: azithromycin — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: azithromycin
Drug: escitalopram — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: escitalopram
Drug: sertraline — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: sertraline
Drug: ondansetron — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: ondansetron
Drug: Ciprofloxacin — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Ciprofloxacin
Drug: Doxycycline — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Doxycycline
Drug: Levofloxacin — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Levofloxacin
Drug: Methylphenidate — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Methylphenidate
Drug: Sumatriptan — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Sumatriptan
Drug: Citalopram — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Citalopram
Drug: Cyclobenzaprine — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Cyclobenzaprine
Drug: Furosemide — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Furosemide
Drug: Gabapentin — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Gabapentin
Drug: Hydrochlorothiazide — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Hydrochlorothiazide
Drug: Hydroxyurea — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Hydroxyurea
Drug: Rosuvastatin — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Rosuvastatin
Drug: Topiramate — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Topiramate
Drug: Trazodone — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Trazodone
Drug: Valganciclovir — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Valganciclovir
Drug: Venlafaxine — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Venlafaxine
Drug: Verapamil — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Verapamil
Drug: Remdesivir — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Remdesivir
Drug: Anakinra — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Anakinra
Drug: Tocilizumab — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Tocilizumab
Drug: Fluvoxamine — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Fluvoxamine
Drug: Amoxicillin — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Amoxicillin
Drug: Bupropion — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Bupropion
Drug: Duloxetine — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Duloxetine
Drug: Hydrocodone — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Hydrocodone
Drug: Levetiracetam — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Levetiracetam
Drug: Paroxetine — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Paroxetine
Drug: Buprenorphine — Understudied drugs will be administered in accordance with local SOC as prescribed by the lactating woman's healthcare provider.
  Groups: Buprenorphine

SUMMARY:
Over half of women in the US who are breastfeeding their infants take prescription drugs. You are being asked to participate in this study because you are breastfeeding your infant and are currently taking, as part of your medical care, at least one of the drugs we are studying. We are interested in studying drugs commonly prescribed to women who are breastfeeding so we can learn more about the amount of drug that is transferred to breastmilk and estimate how much of drug that is consumed by breastfed infants.

DETAILED DESCRIPTION:
The purpose of this study is to understand if the study drugs of interest are found in breastmilk and how much; to estimate the amount of drug that is consumed by breastfed infants and what effect this may have on infants; and to share what we learn with other researchers. The study drugs of interest have Food and Drug Administration (FDA) approval, but there is little or no information about the amount of drug found in the breastmilk of mothers who take them; the amount of drug that may be transferred to their infant's through breastmilk; or the effects this transfer may have on their infants. During this study we will ask to collect breastmilk and blood from mothers, and blood from infants, to measure the amount of study drug of interest in these body fluids. Results from this study will help researchers better understand how much of the study drug of interest is in your blood and breastmilk, and how much of the study drug of interest may be in your infant's blood because of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Lactating women who are receiving at least one DOI per SOC who are ≤180 days postpartum, and their infants (≤180 days of age) who receive maternal breastmilk.
* Informed consent/HIPAA obtained, according to local IRB/REB/IEC guidelines, prior to any study-related procedures. Lactating women who are not legal adults and their breastfed infants may be enrolled if they assent to participate in the study and consent is obtained from their legal guardian according to local IRB/REB/IEC guidelines.

Exclusion Criteria:

* Any concomitant condition which, in the opinion of the physicians providing patient care or the principal investigator conducting the study, would preclude a subject's participation in the study.
* Known pregnancy during PK sampling.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lactating women receiving DOIs per SOC, as prescribed by their healthcare providers, and their breastfed infants.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
M/P ratio | Until the infant becomes 180 days of age
  Characterize the pharmacokinetics using maternal milk/plasma exposure ratio is calculated by dividing the BMS01 drug of interest breastmilk concentration by the BMS01 drug of interest in maternal plasma concentration.
DID | Until the infant becomes 180 days of age
  Pharmacokinetics is characterized by estimated daily infant dose-daily infant dose which estimates the quantity of drug delivered to an infant via breastmilk in a given day.
RID | Until the infant becomes 180 days of age
  Pharmacokinetics is characterized by relative infant dose is a method of relating the potential dose of the drug delivered to the infant to the typical therapeutic dose given to the mother.
I/M ratio | Until the infant becomes 180 days of age
  Pharmacokinetics is characterized using infant maternal/exposure ratio. IM ratio is calculated using the average infant plasma concentration of the BMS01 drug of interest and historical value of clearance in infants.

SECONDARY OUTCOMES:
Safety profile of commonly used drugs in infants exposed to drugs in breastmilk | Until the infant becomes 180 days of age
  see Cohort 1-31 for listing of drugs
AE | Up until 180 days of age
  Safety profile of commonly used drugs in infants exposed to drugs in breastmilk is characterized by Adverse Events(AE) which are collected at each time point when the study-specific procedure occurred and up until 1 hour after.
SAE | Up until 180 days of age
  Safety profile of commonly used drugs in infants exposed to drugs in breastmilk is characterized by Serious Adverse Events which are directly related to study procedures and were recorded from participants (infant or mother) at each time point when the study-specific procedure occurred and up until 1 hour after.
ESI | Until the infant becomes 180 days of age
  Safety profile of commonly used drugs in infants exposed to drugs in breastmilk is characterized by Events of Special Interest(ESI) which include any pre-specified safety event that could be related to BMS01 drug of interest exposure. ESI's are only assessed for infants and only at study visits from the time the BMS01 DOI was initiated in mother and infant began breast milk feeding through the end of the study / infant age ≤ 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Samia Aleem, MD, Principal Investigator — Duke University
Locations (22):
- United States (20):
  - University of California-San Diego Medical Center, La Jolla, California
  - Loma Linda University Health, Loma Linda, California
  - Northwestern University, Chicago, Illinois
  - Ann and Robert H. Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Indiana University Health, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Children's Hospital and Clinics - Minneapolis, Minneapolis, Minnesota
  - University of New Mexico, Health Sciences Center, Albuquerque, New Mexico
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke University Maternal and Fetal Medicine, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania Department of Maternal Fetal Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania
  - Texas Tech University Health Sciences Center School of Medicine., Amarillo, Texas
  - University of Texas Medical Branch - Galveston, Galveston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - The Women's Hospital of Texas, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Canada (2):
  - Lawson Health Research Institute, London, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Job KM, Dallmann A, Parry S, Saade G, Haas DM, Hughes B, Berens P, Chen JY, Fu C, Humphrey K, Hornik C, Balevic S, Zimmerman K, Watt K. Development of a Generic Physiologically-Based Pharmacokinetic Model for Lactation and Prediction of Maternal and Infant Exposure to Ondansetron via Breast Milk. Clin Pharmacol Ther. 2022 May;111(5):1111-1120. doi: 10.1002/cpt.2530. Epub 2022 Mar 5. PMID 35076931